CLINICAL TRIAL: NCT05822544
Title: A Phase 1/1b Study of Single and Multiple Ascending Doses of TLC 6740 in Healthy Subjects, Including Evaluation of Food Effect and Potential Drug-Drug Interactions, and Preliminary Safety and Efficacy in Subjects With Obesity, With or Without Diabetes
Brief Title: Phase 1/1b Study of TLC-6740 in Healthy Subjects and Subjects With Obesity, With or Without Diabetes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OrsoBio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 6740-CL-101
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Healthy Subjects; Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Tirzepatide

STUDY DESIGN:
Intervention Model Description: This study consists of seven parts: Part A (single-ascending dose), Part B (multiple-ascending dose), Part C (adaptive single- and/or multiple-ascending dose), Part D (relative bioavailability of a tablet formulation of TLC-6740), Part E (drug-drug interaction study to determine the effect of TLC-6740 on drug metabolizing enzymes), Part F (multiple dose of TLC-6740 in subjects with obesity with or without type 2 diabetes mellitus), and Part G (multiple dose of TLC-6740 in subjects with obesity receiving tirzepatide).
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Oral Solution (Experimental): Oral solution of TLC-6740
  Interventions: Drug: TLC-6740 Oral Solution; Other: Placebo Oral Solution
- Tablet (Experimental): Tablet formulation of TLC-6740
  Interventions: Drug: TLC-6740 Tablet; Other: Placebo Tablet
- Drug Metabolizing Enzyme (Experimental): Oral dose of omeprazole, voriconazole, itraconazole, or rifampicin
  Interventions: Drug: TLC-6740 Tablet; Drug: Drug Metabolizing Enzyme
- TLC-6740 + Tirzepatide (Experimental): TLC-6740 tablet + subcutaneous injection of tirzepatide
  Interventions: Drug: TLC-6740 Tablet; Drug: Tirzepatide
- Placebo + Tirzepatide (Experimental): TLC-6740 placebo + subcutaneous injection of tirzepatide

INTERVENTIONS:
Drug: TLC-6740 Oral Solution — Oral solution of TLC-6740
  Arms: Oral Solution
Other: Placebo Oral Solution — Placebo-to-match oral solution TLC-6740
  Arms: Oral Solution
Drug: TLC-6740 Tablet — Tablet formulation of TLC-6740
  Arms: Drug Metabolizing Enzyme; TLC-6740 + Tirzepatide; Tablet
Drug: Drug Metabolizing Enzyme — Oral dose of omeprazole, voriconazole, itraconazole, or rifampicin
  Arms: Drug Metabolizing Enzyme
Drug: Tirzepatide — Subcutaneous injection of tirzepatide
  Arms: TLC-6740 + Tirzepatide
Other: Placebo Tablet — Placebo-to-match tablet formulation of TLC-6740
  Arms: Tablet

SUMMARY:
The phase 1 portion of the study is designed to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of TLC-6740 after single- and multiple-ascending doses in healthy subjects. The phase 1b portion of the study is designed to assess the safety, tolerability, and PK of TLC-6740 in subjects with obesity, with or without type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The primary objectives are to assess the safety, tolerability, and plasma PK of TLC-6740 in healthy subjects and subjects with obesity. The exploratory objective is to evaluate the PD of TLC-6740 in healthy subjects and subjects with obesity, with or without type 2 diabetes. This study is comprised of seven parts: Part A (single-ascending dose), Part B (multiple-ascending dose), Part C (adaptive single- and/or multiple-ascending dose), Part D (relative bioavailability of a tablet formulation of TLC-6740), Part E (drug-drug interaction study to determine the effect of TLC-6740 on drug metabolizing enzymes), Part F (multiple dose of TLC-6740 in subjects with obesity with or without type 2 diabetes mellitus), and Part G (multiple dose of TLC-6740 in subjects with obesity receiving tirzepatide). Up to 48, 50, 100, 8, and 28 healthy subjects will be recruited in Parts A, B, C, D, and E, respectively. Up to 180 and 150 obese subjects will be recruited in Parts F and G, respectively. The effect of food on TLC-6740 PK will also be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, healthy male or female subject between 18 and 55 years of age, inclusive (Parts A-E); male or female subject between 18 and 70 years of age, inclusive (Parts F, G)
* Body mass index (BMI) from 19 to 35 kg/m2, inclusive (Parts A-E); BMI ≥ 30 kg/m2 and ≤ 50 kg/m2 (Parts F, G)
* Estimated glomerular filtration rate (eGFR) ≥ 80 mL/min (Parts A-E); eGFR ≥ 60 mL/min/1.73m2 or eGFR ≥ 45 mL/min/1.73m2, depending on cohort (Parts F, G)
* ALT/AST/ALP ≤ 1 x ULN (Parts A-E); ALT/AST < 3 x ULN, ALP < 1.5 x ULN (Parts F, G)
* Screening laboratory evaluations (hematology, chemistry, and urinalysis) must fall within the normal range of the local laboratory's reference ranges unless the results have been determined by the investigator to have no clinical significance (Parts A-E)
* Subject must have either a normal 12-lead electrocardiogram (ECG) or one with abnormalities that are considered clinically insignificant by the investigator
* Females of childbearing potential must have a negative pregnancy test at Screening and clinic admission
* Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception
* Must, in the opinion of the investigator, be in good health based upon medical history and physical examination, including vital signs

Exclusion Criteria:

* Pregnant or lactating subjects
* Unstable type 2 diabetes (as defined as: HbA1c > 10.0%; treatment with insulin and/or pioglitazone within 90 days prior to Screening; any history of diabetic ketoacidosis, hyperosmolar state, and/or acutely decompensated blood glucose control; hypoglycemia unawareness, hospitalization due to hypoglycemia, or history of severe hypoglycemia [requiring outside assistance to regain normal neurologic status]) (Part F)
* History of type 2 diabetes diagnosed prior
* Medical history of type 1 diabetes or latent autoimmune diabetes of adults (LADA)
* Obesity induced by other endocrinologic disorders (e.g., Cushing syndrome) or diagnosed monogenetic or syndromic forms of obesity (e.g., melanocortin 4 receptor deficiency or Prader-Willi syndrome)
* Known serious hypersensitivity to tirzepatide or any of the excipients in tirzepatide (Part G)
* Subjects who have any serious or active medical or psychiatric illness (including depression) that, in the opinion of the investigator, would interfere with the subject's treatment, assessment, or compliance with the protocol
* Subjects who have received any investigational compound within 30 days or 5 half-lives, whichever is longer, prior to study drug dosing
* Current alcohol abuse that is judged by the investigator to potentially interfere with the subject's compliance or safety
* Current substance abuse that is judged by the investigator to potentially interfere with the subject's compliance or safety
* A positive test result for human immunodeficiency virus (HIV-1) antibody, hepatitis B (HBV) surface antigen, or hepatitis C (HCV) antibody
* Medical history of drug sensitivity or drug allergy (such as anaphylaxis or hepatoxicity)
* Presence or history of cardiovascular disease, including significant cardiovascular disease (including a history of myocardial infarction based on ECG and/or clinical history), history of cardiac conduction abnormalities (including any history of ventricular tachycardia), congestive heart failure, cardiomyopathy with left ventricular ejection fraction < 40%, a family history of Long QT Syndrome, or unexplained death in an otherwise healthy individual between the ages of 1 and 30 years
* Syncope, palpitations, or unexplained dizziness
* Implanted defibrillator or pacemaker
* Medical history of liver disease, including but not limited to alcoholic liver disease, autoimmune disorders (e.g., primary biliary cholangitis, primary sclerosing cholangitis, autoimmune hepatitis), drug-induced hepatotoxicity, Wilson disease, clinically significant iron overload, or alpha-1-antitrypsin deficiency)
* Severe peptic ulcer disease, gastroesophageal reflux disease, or other gastric acid hypersecretory conditions
* History of medical or surgical treatment that permanently alters intestinal absorption (e.g., gastric or intestinal surgery)
* Subjects who have received vaccination for COVID-19 within 14 days of Admission

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 564 (Estimated)
Dates: Start 2023-04-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of TLC-6740 treatment-emergent adverse events | Through study completion: up to Day 15 (Parts A, C); Day 24 (Parts B, C); Day 22 (Part D); Day 49 (Part E); Day 168 (Parts F, G) of the study
  Adverse events (AEs) - severity of the AEs will be graded using the Common Terminology Criteria for AE (CTCAE) (v5.0). The relationship between AEs and the study drug will be indicated as related or not related.
PK of TLC-6740 AUC | Through study completion: up to Day 15 (Parts A, C); Day 24 (Parts B, C); Day 22 (Part D); Day 49 (Part E); Day 168 (Parts F, G) of the study
  Area under the concentration-time curve
PK of TLC-6740 Cmax | Through study completion: up to Day 15 (Parts A, C); Day 24 (Parts B, C); Day 22 (Part D); Day 49 (Part E); Day 168 (Parts F, G) of the study
  Maximum plasma concentration
PK of TLC-6740 tmax | Through study completion: up to Day 15 (Parts A, C); Day 24 (Parts B, C); Day 22 (Part D); Day 49 (Part E); Day 168 (Parts F, G) of the study
  Time to reach Cmax
PK of TLC-6740 t1/2 | Through study completion: up to Day 15 (Parts A, C); Day 24 (Parts B, C); Day 22 (Part D); Day 49 (Part E); Day 168 (Parts F, G) of the study
  Half-life
PK of TLC-6740 CL/F | Through study completion: up to Day 15 (Parts A, C); Day 24 (Parts B, C); Day 22 (Part D); Day 49 (Part E); Day 168 (Parts F, G) of the study
  Apparent clearance, calculated as dose/AUC0-inf

CONTACTS AND LOCATIONS:
Overall Officials: OrsoBio Study Director, Study Director — OrsoBio, Inc
Locations (4):
- New Zealand (4):
  - OrsoBio Auckland Research Site 1, Auckland
  - OrsoBio Auckland Research Site 2, Auckland
  - OrsoBio Auckland Research Site 3, Auckland
  - OrsoBio Research Site, Christchurch